CLINICAL TRIAL: NCT06745778
Title: Evolution of Intracardiac Electrograms Recorded by Left Bundle Branch Pacing Lead in Patients With ICD or CRT-D
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: LBBP-ICD study
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-12

CONDITIONS: Ventricular Tachycardia (VT); Ventricular Fibrillation
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICD or CRT-D patients who have received LBBP implantation: Patients' EGMs can be recorded by Holter DR220

SUMMARY:
The goal of this observational study is to investigate the changes of LBB EGM during daily activities and overdrive pacing at the time of peri-implantation and up to 6-month follow-ups of ICD/CRT-D patients. The main question it aims to answer is:

• Does the LBBP lead can provide accurate, stable, and valid EGM for ICD/CRT-D sensing and detection of ventricular tachyarrhythmia events? In each patient intracardiac EGMs of LBBP lead will be collected by ambulatory Holter monitor at the time of peri-implantation and up to 6-month follow-up. EGM collection will be collected at resting and walking conditions and overdrive pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >=18 yrs.
* Patients indicated for ICD or CRT-D (primary or secondary prevention)
* Patients who recently (<=30 days) received ICD/CRT-D implantation with LBBP
* Patients' EGM can be digitally recorded
* Patients are willing to participate in the study and provide signed informed consent

Exclusion Criteria:

* Patients received CIED upgrade or replacement with old pacing leads
* Patients are pregnant
* Patients participate in another study that will confound this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study selected two study site in China. One is a Tertiary A hospital in Zhejiang Province, and another is a hospital in Shanghai. Both of the two sites locate in south east of China. This study will enroll around 50 subjects who meet the inclusion and exclusion criteria from the ICD or CRT-D patients who have received LBBAP in the two hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
R-wave amplitude of LBB EGM | At the enrollment, 3 months after enrollment and 6 months after enrollment
  Amplitude in millivolt

SECONDARY OUTCOMES:
EGM morphology-LVAT | At the enrollment, 3 months after enrollment and 6 months after enrollment
  LVAT in millisecond, calculated based on electrogram recorded by LBB lead

OTHER OUTCOMES:
echocardiography results-LVEF | At the enrollment and 6 months after enrollment
  LVEF in percentage
echocardiography results-SV | At the enrollment and 6 months after enrollment
  SV in millilitre
echocardiography results-LVEDV | At the enrollment and 6 months after enrollment
  LVEDV in millilitre
echocardiography results-LVESV | At the enrollment and 6 months after enrollment
  LVESV in millilitre
echocardiography results-LVEDD | At the enrollment and 6 months after enrollment
  LVEDD in millimetre
echocardiography results-LVESD | At the enrollment and 6 months after enrollment
  LVESD in millimetre

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Shanghai Tongren Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ponnusamy SS, Ramalingam V, Ganesan V, Syed T, Kumar M, Mariappan S, Murugan S, Basil W, Vijayaraman P. Left bundle branch pacing-optimized implantable cardioverter-defibrillator (LOT-ICD) for cardiac resynchronization therapy: A pilot study. Heart Rhythm O2. 2022 Dec 16;3(6Part B):723-727. doi: 10.1016/j.hroo.2022.08.004. eCollection 2022 Dec. PMID 36589004